CLINICAL TRIAL: NCT01503866
Title: A Phase 1 Study to Investigate the Absorption, Metabolism, and Excretion of [14C]-Bardoxolone Methyl Following a Single Oral Dose Administration in Healthy Male Subjects
Brief Title: A Phase I Study to Investigate the Absorption, Metabolism and Excretion in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 402-C-1003
Record Dates: First submitted 2011-12-22; First posted 2012-01-04 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Healthy
MeSH Terms: interventions — bardoxolone methyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 20 mg bardoxolone methyl (Experimental)
  Interventions: Drug: bardoxolone methyl

INTERVENTIONS:
Drug: bardoxolone methyl — oral, single dose

SUMMARY:
The purpose of this study is to determine the absorption and excretion kinetics of bardoxolone methyl and to determine and characterize metabolites present in plasma, urine and feces in men following a single oral does or 20 mg of [14C]-bardoxolone methyl.

ELIGIBILITY:
Inclusion Criteria:

* Males, between ages 18 and 45 years, inclusive;
* Males will either be sterile or agree to use from Check-in (Day -1) until 45 days following Clinic Discharge, i of the following approved methods of contraception: a male condom with spermicide; a sterile sexual partner; use by female sexual partner of an intrauterine device with spermicide; a female condom with spermicide; contraceptive sponge with spermicide; an intravaginal system (eg, NuvaRing); a diaphragm with spermicide;a cervical cap with spermicide; oral, implantable, transdermal, or injectable contraceptives;
* Within a BMI range 19 to 31 kg/m2, inclusive;
* Willing and able to give written informed consent for study participation and provide consent for access to medical data according to appropriate local data protection legislation, allowing authorization to access medical records that describe events captured in the endpoints;
* Willing and able to cooperate with all aspects of the protocol;
* at least 1 regular bowel movement per day.

Exclusion Criteria:

* Participated in another clinical trial of an investigational drug (or a medical device) within 30 days prior to study entry, or are currently participating in another trial of an investigational drug (or a medical device);
* Participated in a [14C]-study within the last 6 months prior to Check-in (Day -1) for this study. The total exposure from this and any previous study must be within the recommended levels considered safe (per 21 Code of Federal Regulations [CFR] 361.1 2010), for example, less than 5,000 mrem/year whole body exposure;
* Exposure to significant radiation within 12 months prior to Check-in (Day -1);
* Any condition possibly affecting absorption, distribution, metabolism, or excretion of drugs that may confound the analyses conducted in this study;
* Known hypersensitivity to any component in the formulation of the study drug, bardoxolone methyl;
* Evidence or history of or concurrent clinically significant allergic, hematological, endocrine, immunological, renal, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease that in the judgment of the Investigator could potentially either pose a health risk to the subject during the study or influence the study outcome;
* Evidence of hepatic or biliary dysfunction including elevation of total bilirubin, direct bilirubin, AST, ALT, GGT, lactate dehydrogenase, or alkaline phosphatase levels to greater than the upper limit of normal;
* Positive test results for human immunodeficiency virus type 1 or 2 antibody, hepatitis B surface antigen, or hepatitis C virus antibody at Screening;
* Any medical or dental procedure, no matter how minor, that is planned or anticipated to occur during the conduct of the study;
* History of drug or alcohol abuse or dependence within the last year;
* Any vaccination within 30 days prior to Day 1 and throughout the study;
* Use of or need for any systemic drug(s) including vitamins or herbal preparations within 30 days prior to Day 1 or during the study;
* Use of aspirin, non-steroidal anti-inflammatory drugs (NSAIDs), or acetaminophen within 5 days prior to the ingestion of the study drug; use of aspirin or NSAIDs (but not acetaminophen) will be allowed during confinement for isolated episodes of pain at the discretion of the Investigator;
* Donation or receipt of blood or blood components within 4 weeks prior to Screening;
* Any diagnostic or intervention procedure requiring a contrast agent within the 30 days prior to Screening;
* Sustained systolic blood pressure > 140 mmHg or < 100 mmHg or a diastolic blood pressure > 95 mmHg at Screening or baseline measured after 5 minutes in a sitting position;
* A pulse rate at rest in a sitting position of < 45 bpm or > 100 bpm;
* An abnormal Screening ECG which is interpreted by the Investigator to be clinically significant;
* Used tobacco- or nicotine-containing products (eg, cigarettes, cigars, chewing tobacco, snuff) or products for smoking cessation 2 weeks prior to study drug administration or during confinement to the Clinical Research Unit (CRU);
* Treated with any investigational agent within 30 days before Check-in (Day -1) or 5 half-lives or twice the duration of biological effect of the previous investigational drug (whichever is longer);
* A positive history of drug abuse or positive results for screening test for drug(s) of abuse, ethanol, amphetamines, barbiturates, cocaine, opiates, benzodiazepines, cannabinoids, or urine cotinine (indicating active current smoking) at the Screening or Check-in (Day -1) visits;
* Poor peripheral venous access;
* Deemed by the Investigator to be inappropriate for this study;
* Any concurrent clinical conditions that in the judgment of the Investigator could either potentially pose a health risk to the subject while involved in the study or could potentially influence the study's outcome.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2011-12-31 (Actual)

PRIMARY OUTCOMES:
area under curve | 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 18, 24, 36, 48, 72, 96, and 120 hours after dose administration

SECONDARY OUTCOMES:
radioactivity in plasma | 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 18, 24, 36, 48, 72, 96, and 120 hours after dose administration
metabolites of ]14C]-bardoxolone methyl | 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 18, 24, 36, 48, 72, 96, and 120 hours after dose administration
Plasma concentrations of cold bardoxolone methyl | 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 18, 24, 36, 48, 72, 96, and 120 hours after dose administration
radioactivity in urine | 0 to 4, 4 to 8, 8 to 12, 12 to 24, 24 to 48, 48 to 72, 72 to 96, 96 to 120,120 to 144, 144 to 168, 168 to 192, 192 to 216, 216 to 240, 240 to 264, 264 to 288, and 288 to 312 hours after dose administration
radioactivity in feces | 0 to 4, 4 to 8, 8 to 12, 12 to 24, 24 to 48, 48 to 72, 72 to 96, 96 to 120,120 to 144, 144 to 168, 168 to 192, 192 to 216, 216 to 240, 240 to 264, 264 to 288, and 288 to 312 hours after dose administration
radioactivity in whole blood | 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 18, 24, 36, 48, 72, 96, and 120 hours after dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Christine L Hale, MD, Principal Investigator — Covance Clinical Research Unit
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/